CLINICAL TRIAL: NCT07149480
Title: Comparison of Postoperative Outcomes of Interlay vs Underlay Graft in Tympanoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaikh Zayed Hospital, Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Israr, Principal Investigator, Shaikh Zayed Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShaikhZayedH1
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Chronic Otitis Media; Tympanic Membrane Perforation; Conductive Hearing Loss
Keywords: Tympanoplasty; Interlay Technique; Underlay Technique; Air-Bone Gap (ABG) Closure; Middle Ear Surgery
MeSH Terms: conditions — Tympanic Membrane Perforation; Hearing Loss, Conductive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Underlay Technique) (Experimental): Patients will undergo tympanoplasty using the underlay graft technique. Under endoscopic guidance, the tympanomeatal flap will be elevated, and the temporalis fascia graft will be placed beneath the remaining tympanic membrane layers along the annulus. The flap will then be repositioned, and the external auditory canal will be packed.
  Interventions: Procedure: Underlay Tympanoplasty
- Group B (Interlay Technique) (Experimental): Patients will undergo tympanoplasty using the interlay graft technique. Under endoscopic guidance, the tympanomeatal flap will be elevated circumferentially. The temporalis fascia graft will be inserted between the fibrous and mucosal layers of the tympanic membrane, particularly beneath the handle of the malleus, before repositioning the flap.
  Interventions: Procedure: Interlay Tympanoplasty

INTERVENTIONS:
Procedure: Underlay Tympanoplasty — Tympanoplasty performed using the underlay graft technique, where the graft is positioned beneath all three layers of the tympanic membrane remnant.
  Other Names: Underlay Graft Placement
  Arms: Group A (Underlay Technique)
Procedure: Interlay Tympanoplasty — Tympanoplasty performed using the interlay graft technique, where the graft is positioned between the mucosal and fibrous layers of the tympanic membrane.
  Other Names: Interlay Graft Placement
  Arms: Group B (Interlay Technique)

SUMMARY:
Chronic otitis media is a long-term ear infection that may cause a hole in the eardrum, leading to repeated ear discharge and hearing loss. When such perforations do not heal on their own, surgery called tympanoplasty is performed to repair the eardrum and improve hearing.

There are different surgical techniques for tympanoplasty. In the underlay technique, the graft (a small piece of tissue used to repair the hole) is placed beneath the layers of the eardrum. This approach is simpler and commonly used, but it carries risks such as displacement of the graft. In the interlay technique, the graft is positioned between specific layers of the eardrum, which may allow more natural healing and better hearing results, but it is technically more demanding.

This clinical study will compare the postoperative outcomes of these two techniques-interlay and underlay-among adults with large central perforations of the eardrum caused by chronic otitis media. The main outcomes assessed will include hearing improvement (measured by closure of the air-bone gap on hearing tests).

We hypothesize that the placement of the graft significantly influences surgical success and hearing recovery. By comparing interlay versus underlay techniques, the study aims to identify which method provides better results for patients. The findings may help refine surgical approaches and improve the overall quality of life for individuals undergoing tympanoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged l6-60 years, of any gender.
* individuals with chronic otitis media characterized by inactive mucosal disease (absence of discharge) accompanied by a large central perforation persisting for at least 6 weeks and exhibiting pure conductive hearing loss as established through pure-tone audiometry.

Exclusion Criteria:

* Presence of active otitis media manifesting acute infection or discharge.
* Patients diagnosed with tympanosclerosis or ossicular necrosis, adversely affecting ossicular chain mobility, as identified in preoperative assessments.
* History of ear surgeries, excluding myringotomy, that could potentially impact tympanoplasty outcomes, such as ossiculoplasty or mastoidectomy.
* Individuals with sensorineural or mixed hearing loss, as determined by pure-tone audiometry, indicating a possible alternate or additional source of hearing impairment.
* Conditions potentially hindering wound healing or compliance with postoperative care, including but not limited to uncontrolled diabetes mellitus or immunodeficiency disorders.
* Patients exhibiting eustachian tube dysfunction, as confirmed through clinical evaluation or medical records.
* Patients with an active focus of infection in the throat, nose, paranasal sinuses, or oral cavity, as determined by medical records.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Mean Hearing Gain (Closure in Air-Bone Gap) | 3 months after surgery
  The average improvement in hearing thresholds, measured by pure-tone audiometry at 500 Hz, 1000 Hz, 2000 Hz, and 4000 Hz. The outcome will be assessed by calculating the difference between the preoperative and postoperative air-bone gap (ABG) values in decibels (dB). This measure evaluates the effectiveness of tympanoplasty in restoring conductive hearing loss.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaikh Zayed Medical college/hospital, Lahore, Lahore, Punjab Province, Pakistan